CLINICAL TRIAL: NCT05648890
Title: Postoperative Cognitive Dysfunction as Geriatric Syndrome
Status: Completed | Type: Observational
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Principal Investigator, Klára Nekvindová, MUDr. Klára Nekvindová - Principal Investigator, Tomas Bata Hospital, Czech Republic
Other Study IDs: ThomasBH
Record Dates: First submitted 2022-11-16; First posted 2022-12-13 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Dysfunction
Keywords: anesthesia, elderly people; PND; POCD; surgery
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients above 65 years old undergoing surgery in general or regional anesthesia.

SUMMARY:
This study is testing cognitive function before and after the surgery, with patient's informed consent. Patients of interest are 65 year or older, undergoing surgery in general or regional anesthesia.

Investigators are using 3 tests. These are: MMSE (Mini Mental State Exam), TEGEST test (test of gestures) and Clock drawing test.

Tests after surgery are performed 2 days until discharge. The testing is anonymous, patient is assigned a number. Main aim of this study is to find a suitable quick test of cognitive function for clinical practice before surgery in general or regional anesthesia.

DETAILED DESCRIPTION:
This study is testing cognitive function before and after the surgery, with patient's informed consent. Patients of interest are 65 year or older, undergoing surgery in general or regional anesthesia.

Investigators are using 3 tests, MMSE - Mini Mental state exam, TEGEST - test of gestures and Clock drawing test with Baja scoring system.

MMSE is 30-point questionnaire. Maximum score for MMSE is 30 points. Score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment. Score 21-23 indicate light cognitive impairment, score 20 - 11 indicate modern cognitive impairment, score 10 points or below indicate severe cognitive impairment.

Maximum score for TEGEST test is 6 points. Score of 4 or less indicates possible cognitive impairments. Patient is showed 6 gestures symbolizing senses (putting on glasses, smelling the flower, looking through telescope, eating with spoon, touching the cheek and picking up the telephone). After showing patient repeats 6 gestures.

Clock drawing test with Baja scoring system is a test, where patient is drawing clock with time 11:10 am. Administrator evaluates 12 digits in the clock, hour hands and pointing of the hour hands. Maximum score for Clock drawing test with Baja scoring system is 5 points. Score 4 or less indicates possible cognitive impairments.

Before testing doctor is assessing Clinical frailty scale (CFS). CSF is tool that can be used to quickly and simply assess frailty. The testing takes place in anesthesiology ambulance before surgery, after operation in clinical wards.

Patients can ask anytime for their results (before or after surgery). A score from 1 (very fit) to 9 (terminally ill) is given based on the descriptions and pictographs of activity and functional status.

Tests after surgery are performed 2 days until discharge. The testing is anonymous a number is assigned to a patients. Patients can refuse anytime to participate in the testing.

The anesthesiologist performing tests is a doctor and can't participate in patient's care in the operating room.

Main aim of this study is to find a suitable quick test of cognitive function for clinical practice before surgery for patients undergoing general or regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older
* absence of sensory impairment (deafness)
* full legal capacity
* informed consent
* ability to speak
* elective or acute surgical procedure

Exclusion Criteria:

* somnolence, coma
* sepsis
* Glasgow coma scale 14 and less
* known psychiatric disease
* effect of premedication, drugs

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients 65 years old and older undergoing surgical procedure in general or regional anesthesia or analgosedation.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ThomasBH, Zlín, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: outcomes of pilot study - 2021 — https://www.prolekare.cz/casopisy/geriatrie-gerontologie/2021-4-23/mereni-perioperacni-neurokognitivni-dysfunkce-u-senioru-nad-65-let-pilotni-studie-129427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were selected by two doctors, main administrator and the colleague. The decision to ask patient about possible enrolment was made 24 hours before preoperative anaesthesiology exam with evaluating online organizer of anaesthesiology outpatient clinic.
Pre-assignment Details: A total of 203 patients participated in the study. A total of 322 potential patients were approached, 268 were screened, 58 were excluded, and 210 were suitable for testing. There were 203 patients who agreed to be included in the study, 39 patients were excluded . The study was completed by 164 patients, whose results were analysed.
Groups:
- Postoperative Cognitive Dysfunction: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Period: Overall Study
Arm/Group | Postoperative Cognitive Dysfunction
Started | 203
Completed | 164
Not Completed | 39

BASELINE CHARACTERISTICS:
Population: Respondents underwent elective, semi-elective or acute surgery under general or regional anaesthesia (orthopaedics and traumatology, general and vascular surgery, neurosurgery, gynaecology, otorhinolaryngology, urology, eye surgery). Preoperative and postoperative testing took place in the anaesthesiology outpatient clinic or at hospital ward.
Groups:
- Group 1 - Postoperative Cognitive Dysfunction as Geriatric Syndrome: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Arm/Group | Group 1 - Postoperative Cognitive Dysfunction as Geriatric Syndrome
Number analyzed (Participants) | 164
Age, Continuous [Median (Standard Deviation); unit: years] | 72 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants] — Respondents underwent elective, semi-elective or acute surgery under general or regional anaesthesia (orthopaedics and traumatology, general and vascular surgery, neurosurgery, gynaecology, otorhinolaryngology, urology, eye surgery). Preoperative and postoperative testing took place in the anaesthesiology outpatient clinic or at hospital ward.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 164
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 164

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Cognitive Dysfunction - Results of MMSE Before Operation
Description: MMSE test was used by administrator before surgery. MMSE is 30 point questionnaire. Maximum score is 30 points. Score of 25 or higher is classed as normal cognitive capacity, 24 points and below is indicating possible congnitive impairment, 21-23 points are light cognitive impairment, 20-11 points are modern impairment, score 10 points or below indicate severe cognitive impairment. The test took 10 minutes approximately.
Time Frame: 2 days before operation
Population: Results of MMSE before operation, descriptive statistics.
Measure: Count of Participants; unit: Participants
Groups:
- Results of MMSE: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Arm/Group | Results of MMSE
Number analyzed (Participants) | 164
Participants
  normal cognitive capacity before operation | 79
  light cognitive impairment before operation | 43
  modern impairment before operation | 37
  severe cognitive impairment before operation | 5
Statistical Analysis 1: Comparison: Results of MMSE; Correlation between MMSE and TEGEST test before operation; Test type: Other — Spearman's rank correlation coefficient was used; p < 0.0001, Spearman's rank correlation coefficient

2. Primary Outcome: Postoperative Cognitive Dysfunction - Results of MMSE After Operation
Description: MMSE test was used by administrator after surgery. MMSE is 30 point questionnaire. Score 25 or higher is know as normal cognitive capacity. Score 24 and below is indicating possible cognitive impairment, score 23-21 points are light cognitive impairment, 20-11 points are mild cognitive impairment, score 10 point or below indicate severe cognitive impairment. The test took 10 minutes approximately.
Time Frame: 3rd day after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Cognitive Dysfunction
Number analyzed (Participants) | 164
Participants
  normal cognitive capacity | 77
  light cognitive impairment | 43
  modern impairment | 38
  severe cognitive impairment | 6
Statistical Analysis 1: Comparison: Postoperative Cognitive Dysfunction; Correlation between MMSE and TEGEST after operation; Test type: Other — Spearman's ran correlation coefficient was used; p < .001, Spearman's ran correlation coefficient; Spearman's ran correlation coefficient was used for correlation between two quantities

3. Primary Outcome: Postoperative Cognitive Dysfunction - TEGEST Test Before Operation
Description: TEGEST test is used by administrator before surgery. Patient is showed 6 gestures symbolizing senses (putting on glasses, smelling the flower, looking through telescope, eating with spoon, touching the cheek, and picking up the telephone). After showing the patient repeats 6 gestures. Maximum score is 6 points, score of 4 or less indicates possible cognitive impairments.
  At the end of testing before surgery administrator did access if patient has possible cognitive impairment. The test took 3 minutes.
Time Frame: 2 days before operation
Population: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Measure: Count of Participants; unit: Participants
Groups:
- TEGEST TEST: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Arm/Group | TEGEST TEST
Number analyzed (Participants) | 164
Participants
  normal cognition | 40
  impairment | 124
Statistical Analysis 1: Comparison: TEGEST TEST; Correlation between TEGEST and Clock drawing test before operation; Test type: Other — Spearman's rank correlation coefficient was used; p < 0.0001, Spearman's rank correlation coefficient; Spearman's rank correlation coefficient was used

4. Primary Outcome: Postoperative Cognitive Dysfunction - TEGEST Test After Operation
Description: TEGEST test is used by administrator after surgery. Patient is showed 6 gestures symbolizing senses (putting on glasses, smelling the flower, looking through telescope, eating with spoon, touching the cheek, and picking up the telephone). After showing the patient repeats 6 gestures. Maximum score is 6 points, score of 4 or less indicates possible cognitive impairments.
  At the end of testing before surgery administrator did access if patient has possible cognitive impairment. The test took 3 minutes.
Time Frame: 3rd day after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Cognitive Dysfunction
Number analyzed (Participants) | 164
Participants
  normal cognition | 77
  cognitive impairment | 87
Statistical Analysis 1: Comparison: Postoperative Cognitive Dysfunction; Correlation between TEGEST and clock drawing test after operation; Test type: Other — Spearman's rank correlation coefficient was used; p < 0.001, Spearman's rank correlation coefficient

5. Primary Outcome: Postoperative Cognitive Dysfunction -Clock Drawing Test Before Operation
Description: Clock drawing test with Baja scoring system is a test, where patient is drawing clock with time given by administrator, which is 11:10 am. Administrator evaluates 12 digits in the clock, hour hands and pointing of the hour hands. Maximum score for is 5 points. Score 4 or less indicates possible cognitive impairment. The test took 3 minutes.
Time Frame: 2 days before operation
Population: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Measure: Count of Participants; unit: Participants
Groups:
- Clock Drawing Test: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Arm/Group | Clock Drawing Test
Number analyzed (Participants) | 164
Participants
  normal cognition | 21
  impairment | 143
Statistical Analysis 1: Comparison: Clock Drawing Test; Correlation between MMSE and Clock drawing test before operation; Test type: Other — Spearman's rank correlation coefficient; p < 0.001, Spearman's rank correlation coefficien
Statistical Analysis 2: Comparison: Clock Drawing Test; Clock drawing before operation; Test type: Other — Mann-Whitney U test before operation; p = 0.023, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Postoperative Cognitive Dysfunction - Clock Drawing Test After Operation
Description: as for outcome 5
Time Frame: 3rd day after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Cognitive Dysfunction
Number analyzed (Participants) | 164
Participants
  normal cognition | 21
  impairment in cognition | 143
Statistical Analysis 1: Comparison: Postoperative Cognitive Dysfunction; Correlation between Clock drawing test and MMSE after operation; Test type: Other — Spearman's rank correlation coefficient; p < 0.0001, Spearman's rank correlation coefficient

7. Secondary Outcome: Clinical Frailty Scale Before Operation
Description: Measure Description: The Clinical Frailty Scale (version 2, by Rockwood) was used preoperatively to assess functional reserve of the patients.
  1= very fit 2 = fit 3 = managing well 4 = living with very mild frailty 5 = living with mild frailty 6= living with moderate frailty 7= living with severe frailty 8= living with very severe frailty 9= terminally ill
Time Frame: 2 days before operation
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Frailty Scale Before Operation: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Arm/Group | Clinical Frailty Scale Before Operation
Number analyzed (Participants) | 164
Participants
  1= very fit | 9
  2 = fit | 43
  3 = managing well | 24
  4 = living with very mild frailty | 23
  5 = living with mild frailty | 24
  6= living with moderate frailty | 22
  7= living with severe frailty | 14
  8= living with very severe frailty | 5
  9= terminally ill | 0
Statistical Analysis 1: Comparison: Clinical Frailty Scale Before Operation; Correlation of Clinical frailty scale with MMSE before operation; Test type: Other — Spearman's rank correlation coefficient was used; p < 0.0001, Spearman's rank correlation coefficient
Statistical Analysis 2: Comparison: Clinical Frailty Scale Before Operation; Correlation of Clinical frailty scale with TEGEST before operation; Test type: Other — Spearman's rank correlation coefficient was used; p < 0.0001, Spearman's rank correlation coefficient
Statistical Analysis 3: Comparison: Clinical Frailty Scale Before Operation; Correlation of Clinical frailty scale with Clock drawing test before operation; Test type: Other — Spearman's rank correlation coefficient was used; p < 0.0001, Spearman's rank correlation coefficient

8. Secondary Outcome: Social Anamnesis Before Operation- Type of Accommodation
Description: Type of accommodation was assessed before operation, options were: house, apartment or institutional accommodation
Time Frame: 2 days before operation
Measure: Count of Participants; unit: Participants
Groups:
- Social Anamnesis Before Operation: Patients above 65 years old undergoing surgery in general or regional anesthesia.
Arm/Group | Social Anamnesis Before Operation
Number analyzed (Participants) | 164
Participants
  apartment | 100
  house | 40
  institution | 24
Statistical Analysis 1: Comparison: Social Anamnesis Before Operation; Respondents living at a house or in apartment and relationships with Clinical frailty scale; Test type: Other — Mann-Whitney U test; p = .562, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Social Anamnesis During Preanesthesia Exam - Living Situation
Description: Living situation of the patients was assessed before operation. Options were living alone or living with someone (family member)
Time Frame: 2 days before operation
Measure: Count of Participants; unit: Participants
Arm/Group | Social Anamnesis Before Operation
Number analyzed (Participants) | 164
Participants
  living with family | 118
  lviing alone | 46
Statistical Analysis 1: Comparison: Social Anamnesis Before Operation; Respondents living with with family or alone and relationship with Clinical frailty scale; Test type: Other — Mann-Whitney test was used; p = 0.129, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Social Anamnesis - Stairs or Elevator
Description: Respondents living at home with stairs and respondents living at home with an elevator
Time Frame: 2nd day before operation
Measure: Count of Participants; unit: Participants
Arm/Group | Social Anamnesis Before Operation
Number analyzed (Participants) | 164
Participants
  stairs | 53
  elevator | 111
Statistical Analysis 1: Comparison: Social Anamnesis Before Operation; Relationship between respondents living at home with stairs and respondents living at home with an elevator and Clinical frailty scale; Test type: Other — Mann-Whintney test was used; p = 0.019, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Adverse events were not monitored or assessed.
Groups:
- Postoperative Cognitive Dysfunction.: Patients above 65 years old undergoing surgery in general or regional anesthesia.
  Patients with adverse events were excluded from the study. Origin of adverse events were not associated with the testing of cognitive function (study was observational).
  Adverse events were: positive test (PCR or antigen) for SARS-CoV-2, severe pain after operation (defined in Numeric Rating Scale as greater than 7), acute respiratory failure, development of somnolence, septic shock after operation or death.
Arm/Group | Postoperative Cognitive Dysfunction.
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Selection bias was due to the way in which patients were enrolled in the study as part of the pre-anaesthetic examination. The first information about possible cognitive impairment was given to the patients during the pre-anaesthetic examination. This information may have caused patients to feel stressed, anxious or worried, and thus may have influenced the test results. The population was limited by patient selection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT05648890/Prot_SAP_000.pdf